CLINICAL TRIAL: NCT04734249
Title: A Multi-cohort and Controlled Study to Evaluate the Efficacy and Safety of Surufatinib Combined With Chemotherapy as Second-line Treatment of Metastatic Colorectal Cancer
Brief Title: Second-line Surufatinib Combined With Chemotherapy in Advanced CRC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HMPL-012-SPRING-C103(SYLT-020)
Record Dates: First submitted 2021-01-28; First posted 2021-02-02 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Advanced Colorectal Cancer

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Advanced CRC (Experimental): Patients with Advanced CRC were given Surufatinib Combined With Chemotherapy
  Interventions: Drug: Surufatinib(HMPL-012)

INTERVENTIONS:
Drug: Surufatinib(HMPL-012) — 1. Cohort 1:Surufatinib(250mg ,qd,po)+mFOLFOX6/FOLFIRI,14 days for a cycle.The curative effect was evaluated every 4 cycles.
     Cohort 2:Surufatinib(250mg ,qd,po)+FOLFOXIRI,14 days for a cycle.The curative effect was evaluated every 4 cycles.
  2. if the first-line chemotherapy was used FoLFOX ,the second-line is FOLFIRI,or the first-line chemotherapy was used FOLFIRI ,the second-line is FoLFOX.
  3. Second-line Surufatinib Combined With Chemotherapy in Advanced CRC.
  Other Names: Chemotherapy(mFOLFOX6/FOLFIRI,FOLFOXIRI)

SUMMARY:
A phase II, muti-cohort study to assess the efficacy and safety of Surufatinib combined with chemotherapy as a second-line treatment in patients with advanced CRC

DETAILED DESCRIPTION:
This study adopt Simon's two-stage minimax designs method based on the primary endpoint of objective response rates. In each arm, 15 patients were planned for the first stage. If two or more responses were observed, an additional 13 patients were to be accrued for a total of 28 patients. If 7 or more of the 28 patients in an arm achieved an objective response, then that arm was designated worthy of additional investigation.

Surufatinib will be orally administered within 1 hour after breakfast once a day (QD) , Cohort 1 :Surufatinib+mFOLFOX6/FOLFIRI,Cohort 2 :Surufatinib+FOLFOXIRI for every 14-day treatment cycle until disease progression, death, intolerable toxicity or other protocol specified end-of-treatment criteria is met (which comes first).

ELIGIBILITY:
Inclusion Criteria

1. Provision of informed consent prior to any study specific procedures, sampling and analyses.
2. Male or female, age18-75 years.
3. Pathologically confirmed unresectable locally advanced or advanced metastatic colorectal adenocarcinoma .
4. The patient had previously failed standard first-line systemic chemotherapy,Prior adjuvant and neo-adjuvant therapy is permitted (chemotherapy, radiotherapy, investigational agents) if 6 months or more have passed since completion of therapy.
5. A WHO performance status equal to 0-1 with no deterioration over the previous 2 weeks and a minimum life expectancy of 12 weeks.
6. At least 1 lesion that has not previously been irradiated, that has not been chosen for biopsy during the study screening period, and that can be accurately measured at Baseline as ≥ 10 mm in the longest diameter (except lymph nodes, which must have short axis ≥ 15mm) with computerized tomography (CT) or magnetic resonance imaging (MRI), whichever is suitable for accurately repeated measurements. If only one measurable lesion exists, it is acceptable to be used (as a target lesion) as long as it has not been previously irradiated and baseline tumour assessment scans are done at least 14days afar the screening biopsy is performed.
7. Inadequate bone marrow reserve or organ function, as demonstrated by any of the following laboratory values:

   1. Absolute neutrophil count (ANC) ≥1.5×109/L
   2. Platelet count ≥100×109 / L
   3. Hemoglobin≥90 g/L（<9 g/dL）
   4. Alanine aminotransferase ≤2.5 × upper limit of normal (ULN) if no demonstrable liver metastases or ≤ 5 × ULN in the presence of liver metastases.
   5. Aspartate aminotransferase (AST) ≤ 2.5 × ULN if no demonstrable liver metastases or ≤ 5 × ULN in the presence of liver metastases.
   6. Total bilirubin (TBL)≤ 1.5 × ULN if no liver metastases or ≤ 3 × ULN in the presence of documented Gilbert's Syndrome (unconjugated hyperbilirubinemia) or liver metastases.
   7. Creatinine≤ 1.5 × ULN concurrent with creatinine clearance ≤50 mL/min (measured or calculated by the Cockcroft-Gault equation); confirmation of creatinine clearance is only required when creatinine is ≤1.5 × ULN.
8. Females should be using adequate contraceptive measures throughout the study; should not be breastfeeding at the time of screening, during the study and until 3 months after completion of the study; and must have a negative pregnancy test prior to start of dosing if of childbearing potential or must have evidence of non-childbearing potential by fulfilling 1 of the following criteria at Screening:

   1. Postmenopausal defined as age more than 50 years and amenorrheic for at least 12 months following cessation of all exogenous hormonal treatments.
   2. Women under 50 years old would be considered postmenopausal if they have been amenorrheic for 12 months or more, following cessation of exogenous hormonal treatments, and with luteinizing hormone (LH) and follicle-stimulating hormone (FSH) levels in the postmenopausal range for the laboratory.Documentation of irreversible surgical sterilization by hysterectomy, bilateral oophorectomy, or bilateral salpingectomy, but not by tubal ligation. Male patients should be willing to use barrier contraception (i.e., condoms).
   3. For inclusion in study, patient must provide a written informed consent.

Exclusion Criteria:

1. Treatment with any of the following:

   1. Prior treatment with Surufatinib .
   2. Major surgery (excluding placement of vascular access) within 4 weeks of the first dose of study drug.
   3. Radiotherapy with a limited field of radiation for palliation within 4 week of the first dose of study drug, with the exception of patients receiving radiation to > 30% of the bone marrow or with a wide field of radiation within 4 weeks of the first dose of study drug.
2. Patients with other malignancies, except basal cell carcinoma and carcinoma in situ..
3. Any unresolved toxicities from prior therapy greater than Common Terminology Criteria for Adverse Events (CTCAE) Grade 1 at the time of starting study treatment, with the exception of alopecia and Grade 2, prior platinum-therapy related neuropathy.
4. Spinal cord compression or brain metastases unless asymptomatic, stable, and not requiring steroids for at least 2 weeks prior to start of study treatment.
5. Any evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension or active bleeding diatheses, which, in the Investigator's opinion, makes it undesirable for the patient to participate in the trial OR which would jeopardize compliance with the protocol such as active infection. Screening for chronic conditions is not required.
6. Refractory nausea, vomiting, or chronic gastrointestinal diseases, inability to swallow the study drug, or previous significant bowel resection that would preclude adequate absorption of Surufatinib.
7. Any of the following cardiac criteria:

   1. Mean resting corrected QT interval (QTc) > 470 ms obtained from 3 electrocardiograms (ECGs), using the screening clinic's ECG machine and Fridericia's formula for QT interval correction (QTcF).
   2. Any clinically important abnormalities in rhythm, conduction, or morphology of the resting ECG (e.g., complete left bundle branch block, third-degree heart block, second-degree heart block, PR interval > 250 ms).
   3. Any factors that increase the risk of QTc prolongation or risk of arrhythmic events, such as heart failure, hypokalemia, congenital long QT syndrome, family history of long QT syndrome, or unexplained sudden death under 40 years of age in first degree relatives or any concomitant medication known to prolong the QT interval.
   4. Left ventricular ejection fraction (LVEF) ≤ 40%.
8. Past medical history of interstitial lung disease, drug-induced interstitial lung disease, radiation pneumonitis that required steroid treatment, or any evidence of clinically active interstitial lung disease.
9. Women who are breastfeeding or have a positive urine or serum pregnancy test at the Screening Visit.
10. History of hypersensitivity to any active or inactive ingredient of Surufatinib or to drugs with a similar chemical structure or class to Surufatinib.
11. Patients who are allergic to paclitaxel or other drugs prepared with polyoxyethyl castor oil, carboplatin or other platinum containing compounds.

    Patients with contraindications of Chemotherapy .
12. Judgment by the Investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions, and requirements.
13. Any disease or condition that, in the opinion of the Investigator, would compromise the safety of the patient or interfere with study assessments.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2021-03 (Estimated); Primary Completion 2021-03 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | up to 12 months
  CR + PR rate according to the RECIST version 1.1 guidelines.

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | up to 12 months
  To assess the efficacy of Surufatinib Combined With Chemotherapy as second-line therapy to Advanced CRC, patients by assessment of progression free survival (PFS) using Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1).
Overall survival time | up to 36 months
  OS was calculated from the date of pharmacy to death from any cause.
Assess the anti-tumor activity:DCR | up to 12 months
  Disease control rate (DCR):CR + PR + SD rate according to the RECIST version 1.1 guidelines.

CONTACTS AND LOCATIONS:
Overall Officials: Rongbo Lin, Study Director — Fujian Cancer Hospital

IPD SHARING:
Plan to Share IPD: No